CLINICAL TRIAL: NCT03314376
Title: Individualized Prehabilitation Program for Patients on a Waiting List for a Transplant.
Brief Title: Prehabilitation in Patients on a Waiting List for a Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funded
Sponsor: University of Malaga (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREHAB-T
Record Dates: First submitted 2017-10-05; First posted 2017-10-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2018-12

CONDITIONS: Transplant Dysfunction
Keywords: prehabilitation; surgery; exercise program; transplant; postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation program (Experimental): Individualized physiotherapy strength and muscular endurance with aerobic training, led by physiotherapists in groups of 8-10 participants.
  Interventions: Device: Prehabilitation program
- Control group (No Intervention): They will be instructed to continue their current activities and not to increase objectively levels of physical activity performed during the 6-week intervention.

INTERVENTIONS:
Device: Prehabilitation program — The intervention will be an 6-week program of individualized physiotherapy strength and muscular endurance with aerobic training, led by physiotherapists in groups of 8-10 participants. Each program will be individualized based on the evaluations of muscular strength and endurance as well as determination of aerobic-anaerobic zone transition described in previous studies In sessions of one hour 3 times a week. Each session will consist of 30 minutes of exercises performed on land followed by 20 minutes of continuous running in treadmill.
  In week 1 and 2 participants carry out 3 sets of 15 repetitions (reps) to become familiar with the exercises. From week 3 onwards participants will perform 4 sets of 10 reps. If the participant can do more than 12 reps, weight will be increased. All exercises are conducted supervised to ensure proper technique and adequate progression.
  Arms: Prehabilitation program

SUMMARY:
The aim of this study is to prove the effects of a individualized prehabilitation program (muscular strength and endurance) in patients in a waiting list for a transplant. The investigators want to see if patients that did a prehabilitation program have better results in the postoperative period.

DETAILED DESCRIPTION:
Some characteristics of the fragile people, like as sarcopenia, are related with worse results after a transplant. Increasing the cardiorespiratory fitness with an exercise program during the preoperative period has shown improvements in patients after a surgery. It is produced a decreased in his functions, including a loss of muscle mass.

Prehabilitation is a exercise program before a surgery. This program will improve the patient's starting functional status and therefore recovery.

Physical activity is one of the most powerful predictors of mortality risk. Several studies say that a improved cardiorespiratory fitness by exercise before a surgery has a great impact in the patients after the intervention in short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients on a waiting list for a transplant.
* Fried Fragility Index >3
* Space more than 6 week between the beginning of the exercise program and the surgery.

Exclusion Criteria:

* Severe cardiovascular disease.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-02 (Estimated); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative length of stay | 10 min
  Days that the patient is in the hospital after the surgery

SECONDARY OUTCOMES:
SF-12 | 10 min
  The state of physical and mental health. SF-12 is a self-administered instrument with 12 items on physical and mental health status; responses are scored (for intensity or frequency) on a Likert-type scale (3-6 points according to the item). This instrument has shown adequate reliability (ICC = 0.73-0.86).
EuroQoL-5D | 10 min
  Quality of life. An auto-informed questionnaire consists of health problems related to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems or extreme problems. Answers are given related to the day when patient completes the questionnaire.
  A quality of life visual analogue scale or VAS ('Best imaginable health state' (100) and 'Worst imaginable health state' (0)). This instrument has shown adequate reliability (0.86 and 0.90).
Profile of Mood States | 10 min
  It is possible to obtain an overall index of altered mood and seven partial measures: stress / anxiety, depression / rejection, anger / hostility, vigor / activity, fatigue / inertia and confusion / bewilderment
Central Sensitization Inventory | 10 min
  Symptoms related to central sensitization
Self-Efficacy/Social Support Scales for Activity | 10 min
  Social needs for the exercise. 4 dimensions (self-efficacy, family, staff and peers) will be assessed with 6 items per dimension (0-6).
Quadriceps strength | 5 min
  Strength peak of knee extension (quadriceps) by one dynamometry instrumented with Powertruck II of Jtech, following the protocol described by Daniels & Worthingham (1995).
Hamstring strength | 5 min
  Strength peak of knee flexion (hamstring) by one dynamometry instrumented with Powertruck II of Jtech, following the protocol described by Daniels & Worthingham (1995).
Brachial triceps strength | 5 min
  Strength peak of elbow extension (brachial triceps) by one dynamometry instrumented with Powertruck II of Jtech, following the protocol described by Daniels & Worthingham (1995).
Biceps brachii strength | 5 min
  Strength peak of elbow flexion (biceps brachii) by one dynamometry instrumented with Powertruck II of Jtech, following the protocol described by Daniels & Worthingham (1995).
Hand grip strength | 5 min
  Hand grip strength will be evaluated by the hydraulic dynamometer Jamar.
Orthogoniometry | 10 min
  The investigators will assess the mobility of the subject. It will be measured the muscular shortening using goniometry (grades=º).
Biochemical markers (Haemogram) | 10 min
  It will be measured in blood samples following clinical standards in 10 ml venous blood. The markers will be HB (hemoglobin), TLC (total WBC count), RBC count, MCV (mean corpuscular volume), MCH (mean corpuscular hemoglobin), MCHC (mean corpuscular hemoglobin concentration), neutrophils, lymphocytes, monocytes, eosinophils, basophils, PCV (packed cell volume), platelet count, P/S (peripheral smear) examination, RDW-SD (RBC distribution width-standard deviation), RDW-CV (RBC distribution width-coefficient of variation), PDW (platelet distribution width), MPV (mean platelet volume), P-LCR (platelet large cell ratio), PCT (platelet crit), absolute neutrophils count, absolute lymphocytes count, absolute monocytes count, absolute eosinophils count, absolute basophils count, and ESR (erythrocyte sedimentation rate).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Study Director — University of Malaga
Locations (1):
- Malaga, Málaga, Spain

REFERENCES:
- [Background] Arthur HM, Daniels C, McKelvie R, Hirsh J, Rush B. Effect of a preoperative intervention on preoperative and postoperative outcomes in low-risk patients awaiting elective coronary artery bypass graft surgery. A randomized, controlled trial. Ann Intern Med. 2000 Aug 15;133(4):253-62. doi: 10.7326/0003-4819-133-4-200008150-00007. PMID 10929164
- [Background] Bao Y, Dalrymple L, Chertow GM, Kaysen GA, Johansen KL. Frailty, dialysis initiation, and mortality in end-stage renal disease. Arch Intern Med. 2012 Jul 23;172(14):1071-7. doi: 10.1001/archinternmed.2012.3020. PMID 22733312
- [Background] Levett DZ, Grocott MP. Cardiopulmonary exercise testing, prehabilitation, and Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):131-42. doi: 10.1007/s12630-014-0307-6. Epub 2015 Jan 22. PMID 25608638
- [Background] Santa Mina D, Clarke H, Ritvo P, Leung YW, Matthew AG, Katz J, Trachtenberg J, Alibhai SM. Effect of total-body prehabilitation on postoperative outcomes: a systematic review and meta-analysis. Physiotherapy. 2014 Sep;100(3):196-207. doi: 10.1016/j.physio.2013.08.008. Epub 2013 Nov 13. PMID 24439570
- [Background] Smith TB, Stonell C, Purkayastha S, Paraskevas P. Cardiopulmonary exercise testing as a risk assessment method in non cardio-pulmonary surgery: a systematic review. Anaesthesia. 2009 Aug;64(8):883-93. doi: 10.1111/j.1365-2044.2009.05983.x. PMID 19604193
- [Background] Cuesta-Vargas AI, Adams N, Salazar JA, Belles A, Hazanas S, Arroyo-Morales M. Deep water running and general practice in primary care for non-specific low back pain versus general practice alone: randomized controlled trial. Clin Rheumatol. 2012 Jul;31(7):1073-8. doi: 10.1007/s10067-012-1977-5. Epub 2012 Mar 29. PMID 22453844
- [Background] Cuesta-Vargas AI, Heywood S. Aerobic fitness testing in chronic nonspecific low back pain: a comparison of deep-water running with cycle ergometry. Am J Phys Med Rehabil. 2011 Dec;90(12):1030-5. doi: 10.1097/PHM.0b013e318238a29c. PMID 22019978
- [Background] Karmali KN, Davies P, Taylor F, Beswick A, Martin N, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2014 Jun 25;(6):CD007131. doi: 10.1002/14651858.CD007131.pub3. PMID 24963623